CLINICAL TRIAL: NCT02164266
Title: A Study to Investigate in Healthy Volunteers (Part 1) and in Patients With Type 2 Diabetes Mellitus (Part 2) the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Doses of RO6799477
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP29205; 2014-000718-78 (EudraCT Number)
Record Dates: First submitted 2014-06-06; First posted 2014-06-16 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Healthy Volunteer, Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Part 1: Healthy Volunteers (Experimental)
  Interventions: Drug: Placebo; Drug: RO6799477
- Part 2: Patients with T2D, Group A (Experimental): Low dose daily oral administration of RO6799477
  Interventions: Drug: Placebo; Drug: RO6799477
- Part 2: Patients with T2D, Group B (Experimental): High dose daily oral administration of RO6799477
  Interventions: Drug: Placebo; Drug: RO6799477

INTERVENTIONS:
Drug: Placebo — Matching placebo daily oral administration
Drug: RO6799477 — Daily oral administration of RO6799477

SUMMARY:
This study is designed to investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of RO6799477 following once daily oral administration for 2 weeks in healthy volunteers (Part 1) and in Type 2 diabetes patients (T2D) (Part 2). The anticipated time on study treatment is two weeks.

ELIGIBILITY:
Inclusion Criteria:

Part 1 Inclusion criteria:

* Right-handed male volunteers
* Aged 18-45 years, inclusive
* Healthy participants, as determined by screening assessments and Principal Investigator's judgment
* Healthy status is defined by the absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, serology and urinalysis
* Body Mass Index (BMI) of 18-30 kg/m2 inclusive, with body weight in the range of 50-100 kg

Part 2 Inclusion Criteria:

* Patients with type 2 diabetes according to WHO criteria diagnosed for at least 3 months prior to screening
* Male or female patients, 40 to 65 years of age, inclusive
* Type 2 diabetic patients who are either drug naive (diet & exercise alone) or on a stable dose of metformin for at least 3 months prior to screening or willing to safely stop sulfonylurea medications at least 2 weeks prior to first dose administration and until follow-up visit
* BMI of 23-42 kg/m2, inclusive

Exclusion Criteria:

Part 1 Exclusion criteria:

* Any clinically relevant history or the presence of e.g. respiratory, renal, hepatic, gastrointestinal, hematological, lymphatic, neurological, cardiovascular, psychiatric, etc. disease or diseases
* Disorders of central nervous system, psychiatric disorders, behavioral disturbances (e.g. cerebrovascular events, depression, post-traumatic stress disorder [PTSD], anxiety, bipolar disorder, severe migraine, Parkinson's disease)
* Participation in an investigational drug or device study within 3 months prior to screening or more than 4 times per year
* Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study

Part 2 Exclusion Criteria:

* Type 1 diabetes
* Acquired or secondary forms of diabetes such as those resulting from pancreatic surgery/injury, cystic fibrosis related diabetes
* Evidence or history of clinically significant diabetic complications such as clinically severe diabetic peripheral neuropathy, clinically significant nephropathy as judged by the investigator, or pre-proliferative/proliferative diabetic retinopathy as judged by the investigator or already diagnosed by the diabetologist or general practitioner
* Disorders of central nervous system, psychiatric disorders, behavioral disturbances
* Clinically significant history or presence of bronchopulmonary, gastrointestinal, hematological, lymphatic, neurological, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, infectious, connective tissue or inflammatory diseases, and any type of cancer (with the exception of treated basal cell carcinoma of the skin) or other clinically significant disease
* Use of anti-diabetic drugs other than metformin or sulfonylureas within 2 months prior to screening
* Any condition or disease detected during the medical interview / physical examination that would render the patient unsuitable for the study, place the patient at undue risk or interfere with the ability of the patient to complete the study in the opinion of the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 9 weeks

SECONDARY OUTCOMES:
Pharmacokinetic parameters derived from plasma and urine concentrations of RO6799477, area under the concentration time curve (AUC), Cmax | Day 1 and Day 14
Fasting serum glucose | Up to 9 weeks
Fasting serum insulin (Part 2 only) | Up to 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Leiden, Netherlands